CLINICAL TRIAL: NCT02330718
Title: Prospective and Retrospective Cohort Study to Find New Prognostic Factors and Therapeutic Targets in Patients With Newly Diagnosed or Relapsed Malignant Hematologic Disorder Excluding Acute Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0236
Record Dates: First submitted 2014-12-29; First posted 2015-01-05 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Malignant Hematologic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — peripheral blood and bone marrow aspirates have been collected and stored for the study
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to elucidate the factors which are associated with the diagnosis and predict prognosis and therapeutic targets by collecting specimens of tissue sample, peripheral blood, and bone marrow aspirates at the time of diagnosis or relapse/refractory in patients with malignant hematologic disorders except acute leukemia. This study is eligible for patients who are diagnosed with malignant hematologic disorders except acute leukemia or who will have diagnostic procedure with suspicion of having hematologic malignancy. Prospective cohort is for patients who are not in treatment for hematologic malignancy. Retrospective cohort is for patients who are diagnosed and in treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients with malignant hematologic disorders except acute leukemia who are diagnosed pathologically according to the revised 2008 WHO classification of tumours of haematopoietic and lymphoid tissue or who will have diagnostic procedure with suspicion of having hematologic malignancy.
* Any gender and age ≥ 19 years
* Written informed consent
* Diagnosed after 2005-01-01 in retrospective cohort group.

Exclusion Criteria:

* Patients who cannot understand or disagree the informed consent
* Patients who diagnosed with acute leukemia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed or relapsed malignant hematologic disorders except acute leukemia
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-05; Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
the number of patients with malignant hematologic disorders to examine the new prognostic factors and therapeutic targets | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea